CLINICAL TRIAL: NCT03724656
Title: Effects of Intraoperative Stimulation of Acupoints on Postoperative Gastrointestinal Motility Recovery in Patients Undergoing Non-gastrointestinal Abdominal Surgery: A Multicenter Randomized Controlled Trial
Brief Title: Effects of Intraoperative Stimulation of Acupoints on Postoperative Gastrointestinal Motility Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Department of Anesthesiology, Director, Chief physician, Professor, Doctoral tutor Affiliation: Tianjin Nankai Hospital, Tianjin Nankai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Gastrointestinal RCT
Record Dates: First submitted 2018-10-28; First posted 2018-10-30 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Gastrointestinal Dysfunction
Keywords: Transcutaneous Acupoint Electrical Stimulation; non-gastrointestinal abdominal surgery; gastrointestinal motility
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture treatment (Experimental): Patients in the TAES treatment group received Transcutaneous Acupoint Electrical Stimulation(TAES) 30 minutes before induction of anesthesia. Bilateral Neiguan（PC6）, bilateral Zusanli（ST36）and bilateral Hegu （LI4）point were selected by electroacupuncture stimulation apparatus (HANS G6805-2, Huayi Co, Shanghai, China).After "Deqi", electroacupuncture stimulation apparatus is connected and maintained until the end of operation.
  Interventions: Device: acupuncture treatment
- Sham acupuncture treatment (Sham Comparator): The control group was treated with non-acupoint shallow acupuncture method. The needle was inserted 5 cm beside the acupoint and the needling depth was less than 2 mm. At the same time, the manual stimulation and "Deqi" was avoided.
  Interventions: Device: sham acupuncture treatment

INTERVENTIONS:
Device: acupuncture treatment — TAES treatment 30 minutes before induction of anesthesia. Bilateral Neiguan（PC6）, bilateral Zusanli（ST36）and bilateral Hegu （LI4）point were selected by electroacupuncture stimulation apparatus (HANS G6805-2, Huayi Co, Shanghai, China).After "Deqi", electroacupuncture stimulation apparatus is connected and maintained until the end of operation.
  Arms: acupuncture treatment
Device: sham acupuncture treatment — Participants in the sham acupuncture group received shallow needling (0.30mm×25mm) at bilateral sham points(nonacupoints located 5cm beside acupoints, about 20mm). The control group was treated with non-acupoint shallow acupuncture method and the needling depth was less than 2 mm. At the same time, the manual stimulation and "Deqi" was avoided.
  Arms: Sham acupuncture treatment

SUMMARY:
1. Research name: Effects of intraoperative stimulation of acupoints on postoperative gastrointestinal motility recovery in patients undergoing non-gastrointestinal abdominal surgery.
2. Research center: Multicenter research
3. Research design: A randomized controlled study method would be used in this study, in which the investigators would provide electroacupuncture on the basis of general anesthesia for non-gastrointestinal abdominal surgery. The effects of electroacupuncture on postoperative gastrointestinal motility recovery in patients undergoing non-gastrointestinal abdominal surgery will be observed and compared with the control group.
4. Research population: Patients who are greater or equal to 18 years old and less than 64 years old , meanwhile intend to receive selective/limited non-gastrointestinal surgery under general anesthesia.
5. Number of participants: 600
6. Interventions: The treatment group received electroacupuncture intervention 30 minutes before induction of anesthesia. In the treatment group, bilateral Neiguan point, bilateral Zusanli point and bilateral Hegu point were selected, then electroacupuncture was applied and the needle was retained until the end of operation. The control group was treated with non-acupoint shallow acupuncture method. The needle was inserted 5 cm beside the acupoint and the needling depth was less than 2 mm. At the same time, the manual stimulation was avoided, "Deqi" was not obtained, electroacupuncture was applied, electric current was regulated, and the needle was retained until the end of the operation.

DETAILED DESCRIPTION:
This study is a large sample, randomized, double-blinded, placebo-controlled and long-term follow-up design. In this study, bilateral Neiguan(PC6), bilateral Zusanli(ST36)and bilateral Hegu (LI4)points were selected for perioperative TAES treatment. accompanied with evaluating the postoperative gastrointestinal motility, the incidence of postoperative nausea and vomiting , as well as the effects on postoperative NRS pain and sleep quality scores . To clarify the effect of TAES on the postoperative spontaneous voiding in patients for laparoscopic surgery is of great significance to the clinical applications and popularization of traditional acupuncture treatment perioperatively across the world.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria

Subjects enrolled in this study must accord with all of the following criteria:

1. Age ≥ 18 years old and <64 years old, gender, ethnicity is not limited;
2. It is intended to selective/limited non-gastrointestinal surgery under general anesthesia;
3. Agree to participate in the study and sign an informed consent form;

Exclusion Criteria:

1. Refusing to participate in this study;
2. Patients with cardiac pacemakers and some special groups, such as pregnant women and those who have had many long-term acupuncture treatment experience;
3. Patients with peptic ulcer, perforation or obstruction;
4. Patients with chronic liver and renal dysfunction, and those who use β-blockers or antihypertensive drugs;
5. The attending doctors or researchers believe that there are other unsuitable situations for the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
postoperative venting | an average of 1 year
  Record the time from the end of the procedure to the patient's first venting after operation

SECONDARY OUTCOMES:
Biochemical tests | 12 months
  Plasma motilin，gastrin ，Vasoactive intestinal peptide (VIP)，SOD（Superoxide Dismutase） and MDA（Malonaldehyde）
bowel sounds and defecation | an average of 1 year
  record the recovery time of postoperative bowel sounds and defecation
Postoperative nausea and vomiting | 12 months
  Record the incidence of postoperative nausea and vomiting in patients

CONTACTS AND LOCATIONS:
Overall Officials: Yu Jianbo, Professor, Study Chair — Nankai Hospital of Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee CH, Kim DK, Yook TH, Sasaki M, Kitamura N. Effectiveness of electroacupuncture at Zusanli (ST36) on the immunohistochemical density of enteroendocrine cells related to gastrointestinal function. J Acupunct Meridian Stud. 2012 Apr;5(2):63-71. doi: 10.1016/j.jams.2012.01.002. Epub 2012 Feb 4. PMID 22483184
- [Background] Wang CP, Kao CH, Chen WK, Lo WY, Hsieh CL. A single-blinded, randomized pilot study evaluating effects of electroacupuncture in diabetic patients with symptoms suggestive of gastroparesis. J Altern Complement Med. 2008 Sep;14(7):833-9. doi: 10.1089/acm.2008.0107. PMID 18721079
- [Background] Gungorduk K, Ozdemir IA, Gungorduk O, Gulseren V, Gokcu M, Sanci M. Effects of coffee consumption on gut recovery after surgery of gynecological cancer patients: a randomized controlled trial. Am J Obstet Gynecol. 2017 Feb;216(2):145.e1-145.e7. doi: 10.1016/j.ajog.2016.10.019. Epub 2016 Oct 22. PMID 27780709